CLINICAL TRIAL: NCT03665116
Title: Effects of Arginine on Osteoarthritis: A Pilot Clinical Trial
Brief Title: Effects of Dietary Supplement on Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Ocean Frontier Institute (Unknown)
Responsible Party: Principal Investigator, Guangju Zhai, PhD, Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20190018
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Gene expression; Molecular phenotype; Osteoarthritis severity grading
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arginine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arginine (Experimental): L-arginine 1.5 g capsule by mouth, once daily for 6 months
  Interventions: Dietary Supplement: L-arginine
- No Intervention (No Intervention): no supplement for 6 months

INTERVENTIONS:
Dietary Supplement: L-arginine — L-arginine capsule
  Arms: Arginine

SUMMARY:
This study evaluates the effects arginine on osteoarthritis (OA) in adults. Participants will be randomly divided into two groups, taking arginine and nothing, respectively. Outcomes will be evaluated by lab test results on OA joint cartilage and self-administered questionnaires. The hypothesis is that arginine can slow down or reverse OA.

DETAILED DESCRIPTION:
1. Patients that meet the inclusion criteria will be approached by a member from their care team, details of this study will be explained. Verbal consent to screening will be obtained during this phone interview and recorded in the clinical trial database; patients will be screened for their eligibility, and a clinical visit will be arranged for eligible patients.
2. Consent form and questionnaires that are commonly used to collect general health information and assess OA patients' mental and physical functions (General Questionnaire, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and 36-Item Short Form Health Survey (SF-36)) will be mailed to eligible patients. Patients will read consent form and fill up questionnaires.
3. Eligible patients will be reached by phone by the research assistant at a later date to obtain their verbal consent to further contact regarding participating in the study, and consent status will be recorded in the clinical trial database.
4. Initial clinical visit:

   1. All questions and concerns will be answered by researchers, consent form will be signed by participants, research assistant, and one of the investigators, and participants will be given a copy as record.
   2. Questionnaires (baseline) will be collected.
   3. 6.5 ml of blood sample (baseline) will be collected by a qualified research nurse.
   4. Participants will be randomly divided into 2 groups, each group will receive arginine and instruction or nothing, and will take arginine or nothing for 6 months:

      * Group I (n=50): 1.5 g of L-arginine daily.
      * Group II (n=50): No supplement.
5. Pre-admission clinical vist:

   * WOMAC and SF-36 questionnaires (at 6 months of the trial) will be administered.
   * 6.5 ml of blood sample (at 6 months of the trial) will be collected.
6. During total joint replacement surgery, small pieces of replaced joint cartilage tissue, which are normally thrown away, will be collected.
7. At 6 and 12 months after the surgery, participants will be reached via phone by the research assistant to complete WOMAC and SF-36 questionnaires. A blood requisition form will be mailed to participants after the last phone interview for their next scheduled routine fasting blood work; 4 ml of blood sample will be collected for the study and sent to the clinical trail lab by the blood collection centre.
8. Lab testing will be conducted; all outcome data will be obtained and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing total knee replacement surgery in 6 months due to primary knee OA
* Must be ambulatory
* Must live in 50 kilometers perimeter of St. John's, capital city of Newfoundland and Labrador, Canada

Exclusion Criteria:

* Clinical diagnosis of secondary OA or inflammatory arthritis
* Cod liver oil supplementation within 6 months
* Supplementation containing arginine within 6 months
* Osteoporotic fracture, previous knee surgery or arthroscopy within 6 months
* Use of bisphosphonates within 2 years
* Use of Intra-articular viscosupplementation or platelet rich plasma at any point

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Target Gene Expressions in Osteoarthritic Knee Cartilage after 6 Months of Supplementation | up to 20 months
  After participants have been taking arginine or nothing for 6 months, and cartilage tissue has been obtained during participants' total knee replacement surgery, target gene expressions in cartilage are measured with quantitative polymerase chain reaction (qPCR). Genes include cartilage degradation enzymes - matrix metallopeptidase 13 (MMP13), cathepsin K (CTSK), cathepsin B (CTSB), and cartilage syntheses genes - aggrecan (ACAN) and type II collagen (CTXII).

SECONDARY OUTCOMES:
OA Severity Grade of Osteoarthritic Knee Cartilage after 6 Months of Supplementation | up to 6 months
  After participants have been taking arginine or nothing for 6 months, and cartilage tissue has been obtained during participants' total knee replacement surgery, the Osteoarthritis Research Society International (OARSI) cartilage histopathology assessment protocol is used to grade OA severity of cartilage on a 7-point scale, with grade 0 as normal cartilage, 1 to 4 with articular cartilage changes only, and 5 to 6 involving subchondral bone.
WOMAC to Measure Changes in Joint Pain and Function between baseline and at 6 Months | at baseline and in 6 months
  WOMAC is used to collect data on participants' self reported joint pain intensity (5 items) and functional deficit (17 items) on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, and 0-68 for functional deficit, and total scores for joint pain and functional deficit at 6 months are compared to baseline, respectively.
WOMAC to Measure Changes in Joint Pain and Function between baseline and at 6 Months Post-surgery | at baseline and 6 months post-surgery
  WOMAC is used to collect data on participants' self reported joint pain intensity (5 items) and functional deficit (17 items) on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, and 0-68 for functional deficit, and total scores for joint pain and functional deficit at 6 months post surgery are compared to baseline, respectively.
WOMAC to Measure Changes in Joint Pain and Function between baseline and at 12 Months Post-surgery | at baseline and 12 months post-surgery
  WOMAC is used to collect data on participants' self reported joint pain intensity (5 items) and functional deficit (17 items) on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, and 0-68 for functional deficit, and total scores for joint pain and functional deficit at 12 months post surgery are compared to baseline, respectively.
SF-36 to Measure Changes in Physical and Mental Function between baseline and at 6 Months | at baseline and in 6 months
  SF-36 is used to collect data on self reported mental and physical health state on 8 scales: physical functioning (10 items); role limitations due to physical health (4 items); role limitations due to emotional problems (3 items); energy/fatigue (4 items); emotional well-being (5 items); social functioning (2 items); pain (2 items); general health (5 items); and self reported health change within one year. All 36 scores are recoded according to "Scoring Rules for the RAND 36-Item Health Survey (Version 1.0)", and items in the same scale are averaged together to generate 8 scale scores, each ranging between 0-100, with higher scores representing a more favorable health state. Scores at 6 months are compared to baseline.
SF-36 to Measure Changes in Physical and Mental Function between baseline and at 6 Months Post-surgery | at baseline and 6 months post-surgery
  SF-36 is used to collect data on self reported mental and physical health state on 8 scales: physical functioning (10 items); role limitations due to physical health (4 items); role limitations due to emotional problems (3 items); energy/fatigue (4 items); emotional well-being (5 items); social functioning (2 items); pain (2 items); general health (5 items); and self reported health change within one year. All 36 scores are recoded according to "Scoring Rules for the RAND 36-Item Health Survey (Version 1.0)", and items in the same scale are averaged together to generate 8 scale scores, each ranging between 0-100, with higher scores representing a more favorable health state. Scores at 6 months post-surgery are compared to baseline.
SF-36 to Measure Changes in Physical and Mental Function between baseline and at 12 Months Post-surgery | at baseline and 12 months post-surgery
  SF-36 is used to collect data on self reported mental and physical health state on 8 scales: physical functioning (10 items); role limitations due to physical health (4 items); role limitations due to emotional problems (3 items); energy/fatigue (4 items); emotional well-being (5 items); social functioning (2 items); pain (2 items); general health (5 items); and self reported health change within one year. All 36 scores are recoded according to "Scoring Rules for the RAND 36-Item Health Survey (Version 1.0)", and items in the same scale are averaged together to generate 8 scale scores, each ranging between 0-100, with higher scores representing a more favorable health state. Scores at 12 months post-surgery are compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Guangju Zhai, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Total Joint Assessment Clinic, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Sharif B, Kopec J, Bansback N, Rahman MM, Flanagan WM, Wong H, Fines P, Anis A. Projecting the direct cost burden of osteoarthritis in Canada using a microsimulation model. Osteoarthritis Cartilage. 2015 Oct;23(10):1654-63. doi: 10.1016/j.joca.2015.05.029. Epub 2015 Jun 5. PMID 26050868
- [Background] Guermazi A, Roemer FW, Felson DT, Brandt KD. Motion for debate: osteoarthritis clinical trials have not identified efficacious therapies because traditional imaging outcome measures are inadequate. Arthritis Rheum. 2013 Nov;65(11):2748-58. doi: 10.1002/art.38086. No abstract available. PMID 23861096
- [Background] Grant WB, Schwalfenberg GK, Genuis SJ, Whiting SJ. An estimate of the economic burden and premature deaths due to vitamin D deficiency in Canada. Mol Nutr Food Res. 2010 Aug;54(8):1172-81. doi: 10.1002/mnfr.200900420. PMID 20352622
- [Background] Schwalfenberg G. Not enough vitamin D: health consequences for Canadians. Can Fam Physician. 2007 May;53(5):841-54. PMID 17872747
- [Background] McAlindon TE, Felson DT, Zhang Y, Hannan MT, Aliabadi P, Weissman B, Rush D, Wilson PW, Jacques P. Relation of dietary intake and serum levels of vitamin D to progression of osteoarthritis of the knee among participants in the Framingham Study. Ann Intern Med. 1996 Sep 1;125(5):353-9. doi: 10.7326/0003-4819-125-5-199609010-00001. PMID 8702085
- [Background] Bergink AP, Uitterlinden AG, Van Leeuwen JP, Buurman CJ, Hofman A, Verhaar JA, Pols HA. Vitamin D status, bone mineral density, and the development of radiographic osteoarthritis of the knee: The Rotterdam Study. J Clin Rheumatol. 2009 Aug;15(5):230-7. doi: 10.1097/RHU.0b013e3181b08f20. PMID 19654490
- [Background] Ding C, Cicuttini F, Parameswaran V, Burgess J, Quinn S, Jones G. Serum levels of vitamin D, sunlight exposure, and knee cartilage loss in older adults: the Tasmanian older adult cohort study. Arthritis Rheum. 2009 May;60(5):1381-9. doi: 10.1002/art.24486. PMID 19404958
- [Background] Abu el Maaty MA, Hanafi RS, El Badawy S, Gad MZ. Association of suboptimal 25-hydroxyvitamin D levels with knee osteoarthritis incidence in post-menopausal Egyptian women. Rheumatol Int. 2013 Nov;33(11):2903-7. doi: 10.1007/s00296-012-2551-9. Epub 2012 Nov 4. PMID 23124694
- [Background] Heidari B, Heidari P, Hajian-Tilaki K. Association between serum vitamin D deficiency and knee osteoarthritis. Int Orthop. 2011 Nov;35(11):1627-31. doi: 10.1007/s00264-010-1186-2. Epub 2010 Dec 30. PMID 21191580
- [Background] Sanghi D, Mishra A, Sharma AC, Singh A, Natu SM, Agarwal S, Srivastava RN. Does vitamin D improve osteoarthritis of the knee: a randomized controlled pilot trial. Clin Orthop Relat Res. 2013 Nov;471(11):3556-62. doi: 10.1007/s11999-013-3201-6. Epub 2013 Aug 1. PMID 23904246
- [Background] McAlindon T, LaValley M, Schneider E, Nuite M, Lee JY, Price LL, Lo G, Dawson-Hughes B. Effect of vitamin D supplementation on progression of knee pain and cartilage volume loss in patients with symptomatic osteoarthritis: a randomized controlled trial. JAMA. 2013 Jan 9;309(2):155-62. doi: 10.1001/jama.2012.164487. PMID 23299607
- [Background] Arden NK, Cro S, Sheard S, Dore CJ, Bara A, Tebbs SA, Hunter DJ, James S, Cooper C, O'Neill TW, Macgregor A, Birrell F, Keen R. The effect of vitamin D supplementation on knee osteoarthritis, the VIDEO study: a randomised controlled trial. Osteoarthritis Cartilage. 2016 Nov;24(11):1858-1866. doi: 10.1016/j.joca.2016.05.020. Epub 2016 Jun 2. PMID 27264058
- [Background] Jin X, Jones G, Cicuttini F, Wluka A, Zhu Z, Han W, Antony B, Wang X, Winzenberg T, Blizzard L, Ding C. Effect of Vitamin D Supplementation on Tibial Cartilage Volume and Knee Pain Among Patients With Symptomatic Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2016 Mar 8;315(10):1005-13. doi: 10.1001/jama.2016.1961. PMID 26954409
- [Background] McAlindon TE, Jacques P, Zhang Y, Hannan MT, Aliabadi P, Weissman B, Rush D, Levy D, Felson DT. Do antioxidant micronutrients protect against the development and progression of knee osteoarthritis? Arthritis Rheum. 1996 Apr;39(4):648-56. doi: 10.1002/art.1780390417. PMID 8630116
- [Background] Brand C, Snaddon J, Bailey M, Cicuttini F. Vitamin E is ineffective for symptomatic relief of knee osteoarthritis: a six month double blind, randomised, placebo controlled study. Ann Rheum Dis. 2001 Oct;60(10):946-9. doi: 10.1136/ard.60.10.946. PMID 11557651
- [Background] Wluka AE, Stuckey S, Brand C, Cicuttini FM. Supplementary vitamin E does not affect the loss of cartilage volume in knee osteoarthritis: a 2 year double blind randomized placebo controlled study. J Rheumatol. 2002 Dec;29(12):2585-91. PMID 12465157
- [Background] Morris SM Jr. Recent advances in arginine metabolism: roles and regulation of the arginases. Br J Pharmacol. 2009 Jul;157(6):922-30. doi: 10.1111/j.1476-5381.2009.00278.x. Epub 2009 Jun 5. PMID 19508396
- [Background] Zhang W, Sun G, Likhodii S, Liu M, Aref-Eshghi E, Harper PE, Martin G, Furey A, Green R, Randell E, Rahman P, Zhai G. Metabolomic analysis of human plasma reveals that arginine is depleted in knee osteoarthritis patients. Osteoarthritis Cartilage. 2016 May;24(5):827-34. doi: 10.1016/j.joca.2015.12.004. Epub 2015 Dec 18. PMID 26708258
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Vukic M, Neme A, Seuter S, Saksa N, de Mello VD, Nurmi T, Uusitupa M, Tuomainen TP, Virtanen JK, Carlberg C. Relevance of vitamin D receptor target genes for monitoring the vitamin D responsiveness of primary human cells. PLoS One. 2015 Apr 13;10(4):e0124339. doi: 10.1371/journal.pone.0124339. eCollection 2015. PMID 25875760
- [Background] Aref-Eshghi E, Liu M, Harper PE, Dore J, Martin G, Furey A, Green R, Rahman P, Zhai G. Overexpression of MMP13 in human osteoarthritic cartilage is associated with the SMAD-independent TGF-beta signalling pathway. Arthritis Res Ther. 2015 Sep 23;17(1):264. doi: 10.1186/s13075-015-0788-x. PMID 26395178
- [Background] Pritzker KP, Gay S, Jimenez SA, Ostergaard K, Pelletier JP, Revell PA, Salter D, van den Berg WB. Osteoarthritis cartilage histopathology: grading and staging. Osteoarthritis Cartilage. 2006 Jan;14(1):13-29. doi: 10.1016/j.joca.2005.07.014. Epub 2005 Oct 19. PMID 16242352
- [Background] Perez-Portela R, Riesgo A. Optimizing preservation protocols to extract high-quality RNA from different tissues of echinoderms for next-generation sequencing. Mol Ecol Resour. 2013 Sep;13(5):884-9. doi: 10.1111/1755-0998.12122. Epub 2013 May 20. PMID 23683108
- [Background] Aref-Eshghi E, Liu M, Razavi-Lopez SB, Hirasawa K, Harper PE, Martin G, Furey A, Green R, Sun G, Rahman P, Zhai G. SMAD3 Is Upregulated in Human Osteoarthritic Cartilage Independent of the Promoter DNA Methylation. J Rheumatol. 2016 Feb;43(2):388-94. doi: 10.3899/jrheum.150609. Epub 2015 Dec 15. PMID 26669923
- [Background] Livak KJ, Schmittgen TD. Analysis of relative gene expression data using real-time quantitative PCR and the 2(-Delta Delta C(T)) Method. Methods. 2001 Dec;25(4):402-8. doi: 10.1006/meth.2001.1262. PMID 11846609
- [Background] Zhai G, Dore J, Rahman P. TGF-beta signal transduction pathways and osteoarthritis. Rheumatol Int. 2015 Aug;35(8):1283-92. doi: 10.1007/s00296-015-3251-z. Epub 2015 Mar 15. PMID 25773660
- [Background] Zhang W, Likhodii S, Aref-Eshghi E, Zhang Y, Harper PE, Randell E, Green R, Martin G, Furey A, Sun G, Rahman P, Zhai G. Relationship between blood plasma and synovial fluid metabolite concentrations in patients with osteoarthritis. J Rheumatol. 2015 May;42(5):859-65. doi: 10.3899/jrheum.141252. Epub 2015 Mar 1. PMID 25729031
- [Background] Zhang W, Sun G, Aitken D, Likhodii S, Liu M, Martin G, Furey A, Randell E, Rahman P, Jones G, Zhai G. Lysophosphatidylcholines to phosphatidylcholines ratio predicts advanced knee osteoarthritis. Rheumatology (Oxford). 2016 Sep;55(9):1566-74. doi: 10.1093/rheumatology/kew207. Epub 2016 May 9. PMID 27160277